CLINICAL TRIAL: NCT00651079
Title: A Double-Blind, Parallel, Randomized, Placebo-Controlled, Single and Repeat Dose Escalation First Time in Human Study to Investigate the Safety, Tolerability and Pharmacokinetics of GSK1247303 in Healthy Male and Female Subjects
Brief Title: GSK1247303 First Time in Human Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IGZ111452
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Healthy Subjects
Keywords: GSK1247303,; Integrase,; First Time in Human

INTERVENTIONS:
Drug: GSK1247303

SUMMARY:
To determine safety, tolerability and Pharmacokinetics of GSK1247303

ELIGIBILITY:
Inclusion Criteria:

* The subject is healthy. Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and 12-lead ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 50 years of age.
* A female subject is eligible to participate if she is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant):
* A male is eligible to enter and participate in the study if he is surgically sterile OR if he either agrees to abstain from sexual intercourse with a female partner or agrees to use a condom/spermicide, in addition to having his female partner use another form of contraception as outlined in Section 8.1.
* Body weight >=50 kg (110 lbs.) for men and >= 45 kg (99 lbs) for women and body mass index (BMI) within the range 18.5-31.0 kg/m2 (inclusive).
* A signed and dated written informed consent is obtained from the subject or the subject's legal representative prior to screening.
* Subject must be capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* As a result of the medical interview, physical examination, or screening investigations, the Investigator considers the subject unfit for the study.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting surgery or percutaneous transluminal coronary angioplasty or any clinically significant cardiac disease.
* History/evidence of clinically significant pulmonary disease.
* Has a positive pre-study Hepatitis B surface antigen; positive hepatitis C (HCV) antibody or detectable HCV ribonucleic acid (RNA); or positive HIV-1 antibody result.
* Has a history of regular alcohol consumption averaging >7 drinks/week for women or >14 drinks/week for men within 6 months of the screening visit.

Note: 1 drink is equivalent to 12 g alcohol = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.

* Unwilling to abstain from alcohol for 48 hours prior to the start of dosing until collection of the final pharmacokinetic sample during each treatment period.
* Has a history of regular use of tobacco- or nicotine-containing products within 3 months of the screening visit.
* The subject has a positive pre-study drug and/or alcohol screen.
* Unwilling to refrain from the use of illicit drugs and adhere to other protocol-stated restrictions while participating in the study.
* The subject has received an investigational drug or participated in any other research trial within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
* Participation in the study would result in donation of blood in excess of 500 mL within a 56 day period. Note: This does not include plasma donation.
* History or presence of allergy or intolerance to the study drug or its components or drugs of its class, or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation. In addition, if heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled. Note: "Study" or "investigational" drugs include GSK1247303 or placebo.
* Use of prescription or non-prescription drugs, including antacids, vitamins, herbal and dietary supplements (including St John's Wort and iron supplements) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), or total bilirubin values greater than the upper limit of normal. A single repeat is allowed for eligibility determination.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy should be excluded.
* History of significant renal or hepatic diseases.
* History of Gilbert's syndrome.
* Exclusion Criteria for 24-Hour Screening Holter as per protocol.
* Exclusion criteria for screening ECG as per protocol (a single repeat is allowed for eligibility determination).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
safety (adverse events, laboratory, ECG and vital signs assessments) and plasma pharmacokinetics of single and repeat doses of GSK1247303

SECONDARY OUTCOMES:
Day 10 GSK1247303 AUC(0-t) compared to AUC(0-12) and/or AUC(0-24) on Day 1 to estimate accumulation ratio (R) and GSK1247303 AUC(0-t) on Day 10 compared to AUC on Day 1 to evaluate time invariance following repeat administration of GSK1247303. | day 1 and day 10
Pre-morning dose concentrations (Ct) on Day 2 through 10 to assess the achievement of steady state of GSK1247303 following repeat administration. | Day 2 through 10
GSK1247303 PK parameters: AUC(0-t), AUC(0-t), Cmax, and C12 and/or C24 following single dose administration and AUC(0-t), Ct, Cmin, and Cmax following repeat administration at different doses for the assessment of dose proportionality.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States